CLINICAL TRIAL: NCT00745849
Title: Efficacy of Esomeprazole for Non-Allergic Rhinitis: A Double-blind, Placebo Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dave Khan, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Efficacy Esomeprazole NAR
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Vasomotor Rhinitis
Keywords: non-allergic rhinitis, laryngopharyngeal reflux
MeSH Terms: conditions — Rhinitis, Vasomotor; Common Cold; Laryngopharyngeal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): esomeprazole 40mg po bid
  Interventions: Drug: esomeprazole
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: esomeprazole — 40mg by mouth twice daily
  Other Names: Nexium
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
The purpose of this study was to see if high dose esomeprazole (40mg bid) was effective in treating non-allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* age between 18-80, symptoms of perennial rhinitis, negative epicutaneous skin testing to a panel of common aeroallergens, and ability to speak English

Exclusion Criteria:

* pregnancy or breast-feeding, evidence of positive skin tests to a common aeroallergen, treatment with a proton pump inhibitor within the month prior to enrollment, treatment with any other anti-reflux therapy within the last month on a daily basis or within the last two weeks on an as needed basis, and other gastrointestinal disorders leading to reflux symptoms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Khan, MD, Principal Investigator — Department of Allergy and Immunology, UT Southwestern
Locations (1):
- Clinical Trials Office, Aston Building, UT Southwestern, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from UT Southwestern outpatient clinics as well as through flyers and local advertising
Pre-assignment Details: 43 patients were assigned for randomization after meeting inclusion criteria: age between 18-80, symptoms of perennial rhinitis, negative epicutaneous skin testing to a panel of common aeroallergens, and ability to speak English
Groups:
- Placebo First, Then Esomeprazole: Placebo twice daily for 8 weeks, then two week washout, then Esomeprazole 40mg twice daily for 8 weeks
- Esomeprazole First, Then Placebo: Esomeprazole 40mg twice daily for 8 weeks, then two week washout, then Placebo twice daily for 8 weeks
Period: First Intervention
Arm/Group | Placebo First, Then Esomeprazole | Esomeprazole First, Then Placebo
Started | 21 | 22
Completed | 20 | 20
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Washout Period
Arm/Group | Placebo First, Then Esomeprazole | Esomeprazole First, Then Placebo
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Esomeprazole | Esomeprazole First, Then Placebo
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: 37 patients were included in Data Analysis. Study subjects were randomized to esomeprazole 40mg tablet twice daily or placebo for eight weeks each, with a two week washout crossover period in between treatment arms.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 44.9 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 11
Baseline Reflux Score [Mean (Full Range); unit: units on a scale] — Minimum Score = 0 Maximum Score = 14
  The higher the score, the more baseline reflux symptoms
  units on a scale | 4.8 [0 to 11]
Number of Patients on Intranasal Corticosteroids [Count of Participants; unit: Participants] | 4
Number of Patients on Oral Antihistamines [Count of Participants; unit: Participants] | 9
Number of Patients on Oral Leukotriene Receptor Antagonists [Count of Participants; unit: Participants] | 5
Number of Patients on Intranasal Antihistamines [Count of Participants; unit: Participants] | 1
Number of Patients on Intranasal Anticholinergics [Count of Participants; unit: Participants] | 2
Number of Patients on Oral Decongestants [Count of Participants; unit: Participants] | 4
Number of Patients on Intranasal Decongestants [Count of Participants; unit: Participants] | 2
Number of Patients on Nasal Saline Rinses [Count of Participants; unit: Participants] | 3
Number of Patients on Oral Antacids (none in two weeks prior to enrollment) [Count of Participants; unit: Participants] | 7
Nasal Symptom Score : Sneezing [Mean (Full Range); unit: units on a scale] — (1=None, 7=Unbelievably Severe)
  units on a scale | 2.8 [1 to 7]
Nasal Symptom Score : Runny Nose [Mean (Full Range); unit: units on a scale] — (1=None, 7=Unbelievably Severe)
  units on a scale | 3.8 [1 to 6.5]
Nasal Symptom Score : Congestion [Mean (Full Range); unit: units on a scale] — (1=None, 7=Unbelievably Severe)
  units on a scale | 4.4 [1 to 7]
Nasal Symptom Score : Itchy Nose [Mean (Full Range); unit: units on a scale] — (1=None, 7=Unbelievably Severe)
  units on a scale | 2.9 [1 to 6]
Nasal Symptom Score : Postnasal Drip [Mean (Full Range); unit: units on a scale] — (1=None, 7=Unbelievably Severe)
  units on a scale | 4.4 [1 to 7]
Nasal Symptom Score : Total Nasal Symptoms [Mean (Full Range); unit: units on a scale] — (1=None, 7=Unbelievably Severe)
  units on a scale | 4.8 [1.5 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Total Nasal Symptom Scores
Description: (1=none, 7=unbearably severe) difference in nasal symptom scores for the average of the last two weeks of each treatment arm
Time Frame: Last two weeks of each treatment arm
Population: Each study participant was in both arms of the study since this was a crossover study
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Esomeprazole Arm: esomeprazole: 40mg by mouth twice daily for 8 weeks
- Placebo Arm: placebo twice daily for 8 weeks
Arm/Group | Esomeprazole Arm | Placebo Arm
Number analyzed (Participants) | 37 | 37
score on a scale | 3.0 [1 to 6] | 3.1 [1 to 6]
Statistical Analysis 1: Comparison: Esomeprazole Arm vs Placebo Arm; Test type: Superiority; p = 0.45, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Events Occurring While Subject Was on Placebo: This arm includes all patients in the study, but focuses on the time period when they were on Placebo only.
- Events Occurring While Subject Was on Esomeprazole: This arm includes all patients in the study, but focuses on the time period when they were on Esomeprazole only.
Arm/Group | Events Occurring While Subject Was on Placebo | Events Occurring While Subject Was on Esomeprazole
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
Six patients did not complete the study and may have affected the outcome. Optimal duration for treatment of laryngopharyngeal reflux is unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes